CLINICAL TRIAL: NCT01818388
Title: A Multicenter, Prospective, Single Arm Observational Trial to Assess Intravascular Temperature Management (IVTM) in the Treatment of Cardiac Arrest
Brief Title: COOL-ARREST Pilot Study to Assess Intravascular Temperature Management (IVTM) in the Treatment of Cardiac Arrest
Acronym: COOL-ARREST
Status: Completed | Type: Observational
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Other Study IDs: EDC-1978
Record Dates: First submitted 2013-02-04; First posted 2013-03-26 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-04

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IVTM system, therapeutic hypothermia: Induced therapeutic hypothermia post cardiac arrest
  Interventions: Device: ZOLL Intravascular Temperature Management System (IVTM)

INTERVENTIONS:
Device: ZOLL Intravascular Temperature Management System (IVTM) — Induced therapeutic hypothermia post cardiac arrest.

SUMMARY:
A multicenter prospective single arm interventional trial in hospitals where therapeutic hypothermia is standard practice. This trial will enroll 50 subjects to evaluate the ability of the ZOLL Intravascular Temperature Management (IVTM) System to induce, maintain, and reverse mild therapeutic hypothermia and maintain normothermia post cardiac arrest.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent
2. 18 years of age or older
3. Out-of-hospital witnessed cardiac arrest with any rhythm [Ventricular Fibrillation/Tachycardia (VF/VT), Pulseless Electrical Activity (PEA), or Asystole (AS)] during EMS phase of treatment

   OR:

   Out-of-hospital unwitnessed cardiac arrest with VF upon EMS arrival
4. Lack of meaningful response to verbal commands upon arrival to hospital after suffering non-traumatic cardiac arrest in an out-of-hospital setting
5. Return of spontaneous circulation (ROSC) within 30 minutes of EMS arrival
6. Able to maintain a SBP > 90mmHg for 30 minutes post ROSC without the use of pressors OR with stable dose of pressors (if escalation of pressors is required, patient is not eligible)
7. Undergoing Therapeutic Hypothermia using ZOLL's IVTM System within twelve hours of ROSC BUT should have been initiated as soon as possible

Exclusion Criteria

1. Traumatic cardiac arrest [due to blunt trauma, penetrating injury (e.g., stabbing, gunshot, etc.), burns, exsanguinations, strangulation, smoke inhalation, electrocution, hanging, drowning, etc.]
2. Toxicological etiology (e.g., inhalation of toxic substances, drugs, etc.)
3. Known or suspected pregnancy
4. Do Not Attempt to Resuscitate (DNAR) order in force
5. Ward of the state or prisoner
6. Anatomy, previous surgery or disease state contraindicating femoral venous access
7. Received neuromuscular blocking agents or central nervous system sedatives whose effects have not worn off prior to assessing level of consciousness following ROSC
8. Hypothermia initiated at a transferring facility prior to arrival at the enrolling hospital (excludes pre-hospital IV fluids or cold packs for cooling by EMS)
9. Current Inferior Vena Cava (IVC) filter
10. Known history of acute neurological illness or severe functional disabilities prior to arrest (e.g., seizures, traumatic brain injury, increased intracranial pressures, intracerebral hemorrhage, etc.)
11. Known heparin allergy
12. Known allergy to any adjunctive pharmacologic agent required for induction or maintenance of therapeutic hypothermia
13. Known history of bleeding or blood disorders such as coagulopathy, cryoglobulinemia, sickle cell or thrombocytopenia with a platelet count below 40,000.
14. Known hypersensitivity to hypothermia including a history of Raynaud's disease
15. Evidence of intracranial bleed
16. Terminal illness or life expectancy of less than 3 months prior to arrest
17. Currently enrolled in another investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with this trial's endpoints Note: For the purpose of this protocol, subjects involved in extended follow-up trials for products that were investigational but are currently commercially available are not considered enrolled in an investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have experienced an out-of-hospital cardiac arrest.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in which IVTM can therapeutically cool patients as a measure of Performance | Day 1

SECONDARY OUTCOMES:
Ability to Enroll Subjects, Proportion of those Enrolled that Complete the Study Protocol and Time to complete Enrollment of 50 Subjects Defined as Retention | Up to 90 days
Incident Adverse Events Defined as Safety | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Neil, MD, Principal Investigator — Wayne State University, School of Medicine Specialist and Chief, Detroit Medical Center
Locations (9):
- United States (9):
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Wayne State University / Detriot Medical Center, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Palmetto Health Clinical Trials Department, Columbia, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided